CLINICAL TRIAL: NCT00921102
Title: Intrathecal Atropine to Prevent Nausea and Vomiting After Spinal Anesthesia With Morphine for Elective Caesarean Section: a Randomized Controlled Trial
Brief Title: Atropine to Prevent Nausea and Vomiting After Spinal Anesthesia for Caesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Guido Fanelli, MD, University of Parma
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANEST-OST-01
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Cesarean Section; Anesthesia,Spinal; Postoperative Nausea and Vomiting
Keywords: Atropine; Morphine; Analgesics, Opioid; Antiemetics
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Bupivacaine; Anesthetics, Local; Morphine; Sodium Chloride; Atropine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Patients in this group will receive both an intrathecal and intravenous injection of saline solution, as a placebo comparator.
  Interventions: Drug: Bupivacaine; Drug: Morphine; Drug: Isotonic saline solution
- Intrathecal Atropine (Experimental): Patients in this group will receive intrathecal atropine as a prophylactic antiemetic agent. They will also receive intravenous saline solution to maintain blinding.
  Interventions: Drug: Bupivacaine; Drug: Morphine; Drug: Isotonic saline solution; Drug: Atropine
- IV Atropine (Active Comparator): Patients in this group will receive a small dose of atropine via the intravenous route to examine its possible antiemetic activity. They will also receive intravenous saline solution to maintain blinding.
  Interventions: Drug: Bupivacaine; Drug: Morphine; Drug: Isotonic saline solution; Drug: Atropine

INTERVENTIONS:
Drug: Bupivacaine — 12.5 mg of a 5 mg/ml hyperbaric solution, intrathecally
  Other Names: Local Anesthetic; Hyperbaric Bupivacaine; Marcain Heavy Injection
Drug: Morphine — 200 µg of a 200 µg/ml solution, intrathecally
Drug: Isotonic saline solution — 0.9% NaCl solution
  0.1 ml, intrathecally in group Control and IV Atropine
  0.1 ml, intravenously in group Control and Intrathecal Atropine
  Other Names: Sodium chloride
Drug: Atropine — 100 µg of a 1 mg/ml preservative-free solution
  * intrathecally in group Intrathecal Atropine
  * intravenously in group IV Atropine
  Arms: IV Atropine; Intrathecal Atropine

SUMMARY:
The aim of this study is to assess the efficacy of atropine in preventing nausea and vomiting after spinal anesthesia with local anesthetic and morphine for elective Caesarean section.

Patients enrolling in the study will be assigned to one of three groups. One will receive a small dose of intrathecal atropine; another will receive small-dose intravenous atropine; the third group will receive placebo.

DETAILED DESCRIPTION:
Intrathecal (IT) morphine grants effective, durable and safe analgesia after Caesarean section. The most common adverse effects after IT morphine are widespread pruritus and postoperative nausea and vomiting (PONV).

Postoperative nausea and vomiting is multifactorial in origin; in addition to general and pre-existing risk factors, such as elevated gonadotropin and progesterone serum levels, parturients undergoing Caesarean section are exposed to drug-induced, hemodynamic and surgical (manipulation of the uterus) stimuli.

Anticholinergic agents, and particularly scopolamine, have long been known to decrease opioid-related nausea and vomiting, although their narrow therapeutic range and inconvenient route of administration (typically transdermal) has limited their application. Anticholinergic agents are thought to act via inhibition of muscarinic receptors in several regions of the medulla oblongata, which are implicated with nausea and vomiting generation; in addition to the chemoceptor trigger zone, these receptors are particularly concentrated in, but not limited to the nucleus tractus solitarius. Cholinergic receptors have been typically associated with motion sickness, but cholinergic agonists such as neostigmine have been shown to increase the incidence of PONV, especially when injected intrathecally.

Anticholinergic agents with muscarinic selectivity may be effective in preventing and treating PONV. Intravenous (IV) administration of scopolamine or atropine, but not glycopyrrolate, reduces the incidence of PONV. Intuitively, as glycopyrrolate does not cross the blood-brain barrier, most postoperative anti-emetic effects of anticholinergic drugs should be mediated by central receptors.

Few studies have specifically evaluated the antiemetic effect of IV atropine after balanced general or opioid-based regional anesthesia, with conflicting results. Atropine may represent a valid alternative to scopolamine and its adverse effects; however, its apparent duration of action is "brief" (minutes to 1 hour) when administered IV.

After we became aware of several observations by Ramaioli and De Amici on the efficacy of small-dose intrathecal (IT) atropine for the treatment of PONV after IT morphine administration, we set out to investigate the use of this agent for prophylaxis of PONV in a high-risk population, such as patients receiving IT morphine for postoperative analgesia after elective Caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective Cesarean section at up to 42 weeks and 2 days
* Patients in ASA Physical Status Class I or II
* Informed written consent to participation
* No known gestosis

Exclusion Criteria:

* Any known fetal pathology
* Indication to general anesthesia
* Known allergy to any of the study drugs
* Baseline bradycardia or any cardiovascular disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting (PONV) as expressed by at least one rating > 3 on a numerical rating scale (0-10). | 12 hours post-operatively

SECONDARY OUTCOMES:
Incidence and prevalence of PONV up to 24 h postoperatively, expressed as both ratings on a numerical rating scale and as the area under the curve of these ratings over time. | Up to 24 h postoperatively
Incidence of atropine-related side effects such as xerostomia, anxiety, tachycardia. | Up to 24 h postoperatively
Postoperative pain expressed as time to first request for supplemental analgesia and as rating on a numerical rating scale. | Up to 24 h postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Guido Fanelli, MD, Study Chair — University of Parma; Andrea Cornini, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma, Parma, Italy
Locations (2):
- Italy (2):
  - University of Messina, Messina, ME
  - University and Hospital of Parma (Azienda Ospedaliero-Universitaria di Parma), Parma, PR

REFERENCES:
- [Background] Ramaioli F, De Amici D. Central antiemetic effect of atropine: our personal experience. Can J Anaesth. 1996 Oct;43(10):1079. doi: 10.1007/BF03011915. No abstract available. PMID 8896865
- [Background] Salmenpera M, Kuoppamaki R, Salmenpera A. Do anticholinergic agents affect the occurrence of postanaesthetic nausea? Acta Anaesthesiol Scand. 1992 Jul;36(5):445-8. doi: 10.1111/j.1399-6576.1992.tb03494.x. PMID 1632167
- [Background] Moscovici R, Prego G, Schwartz M, Steinfeld O. Epidural scopolamine administration in preventing nausea after epidural morphine. J Clin Anesth. 1995 Sep;7(6):474-6. doi: 10.1016/0952-8180(95)00056-n. PMID 8534463
- [Background] Kotelko DM, Rottman RL, Wright WC, Stone JJ, Yamashiro AY, Rosenblatt RM. Transdermal scopolamine decreases nausea and vomiting following cesarean section in patients receiving epidural morphine. Anesthesiology. 1989 Nov;71(5):675-8. doi: 10.1097/00000542-198911000-00009. PMID 2817461
- [Derived] Griffiths JD, Gyte GM, Popham PA, Williams K, Paranjothy S, Broughton HK, Brown HC, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2021 May 18;5(5):CD007579. doi: 10.1002/14651858.CD007579.pub3. PMID 34002866